CLINICAL TRIAL: NCT04936724
Title: Evaluation of the New FDA Warning Labels: Does Highlighting Lesser Known Harms of Tobacco Use Increase Attention, Recall and Knowledge of Tobacco Harms for Young Adults?
Brief Title: FDA Cigarette Warning Labels: Eye Tracking Study
Acronym: FLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Andrew Strasser, Associate Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPCC 04021; U54CA229973 (NIH); 843703 (Other: IRB Protocol Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-23 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Smoking, Cigarette
Keywords: Pictorial warning labels; Cigarette smoking; Eye-tracking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: It is a randomized, parallel design experimental study using objective measures and self-report survey. We will recruit 120 daily smokers (60 young adults and 60 adults) to participate in a single-session laboratory-based study. The participants will be assigned to either the lesser-known or well-known PWL group. After completing a baseline questionnaire, the participants will view 4 warning labels in a randomized order from their assigned group followed by a follow-up questionnaire. Primary outcomes will be eye-tracking measures, label recall and recognition, and knowledge of tobacco harms.
Who Masked: Participant
Masking Description: Participants will be informed that they will be viewing cigarette warning labels during the eye-tracking task, but will be unaware of their randomization condition (lesser-known vs well-known harms)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition A (Lesser-known harms) (Experimental): Participants randomized to this condition will view cigarette warning labels highlighting lesser-known harms of tobacco use.
  Interventions: Other: Pictorial Warning Labels
- Condition B (Well-known harms) (Experimental): Participants randomized to this condition will view cigarette warning labels highlighting the well-known harms of tobacco use.
  Interventions: Other: Pictorial Warning Labels

INTERVENTIONS:
Other: Pictorial Warning Labels — Participants will be randomized to one of two conditions and will view 4 pictorial warning labels from the assigned group for an eye-tracking task.

SUMMARY:
The purpose of this study is to examine the effect of cigarette pictorial warning label content (lesser-known vs well-known risks) on visual engagement, recall, and knowledge of tobacco use harms.

DETAILED DESCRIPTION:
This laboratory-based study will aim to enroll 120 current cigarette users to complete a 1-day randomized, parallel design protocol.

The participants will be randomized to one of two conditions, pictorial warning labels (PWLs) with well-known or lesser-known tobacco harms. After completing a baseline questionnaire, the participants will view 4 warning labels from the assigned group and complete a follow-up questionnaire. Eye-tracking will provide data on visual processing of the warning labels and the effect of these labels on knowledge, attitudes, and beliefs about smoking will be supplemented by self-report.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers using only filtered commercially manufactured cigarettes; smoking at least 5 cigarettes daily and smoking for at least last 1 year.
* Participants must physically present a pack of their preferred brand of cigarettes at the lab session to confirm their status as a cigarette smoker.
* Not currently undergoing smoking cessation treatment or planning to quit smoking currently or in the next month.
* Plan to live in the area for the duration of the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined Informed Consent and HIPAA form.
* Able to communicate fluently in English (i.e., speaking, writing, and reading) as determined by the research assistant.

Exclusion Criteria:

* Use of any nicotine-containing products other than cigarettes. Participants reporting isolated use of other nicotine-containing products less than 5 times per month are eligible to participate.
* Not actively trying to quit smoking currently and had not made a quit attempt in the past month.
* Self-report current alcohol consumption that exceeds 25 standard drinks/week.
* Self-report current pregnancy or breastfeeding.
* Any self-reported impairment - visual (colorblindness or impairments such as glass eye), physical, and/or neurological impairments preventing the proper completion of the study procedures.
* Serious or unstable medical condition.
* Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.
* Current use or discontinuation of anti-psychotic medications within the last 6 months.
* Current diagnosis of active major depression. Participants who maintain a diagnosis of major depression who have not experienced any major depressive episodes in the past 6 months and are stable on antidepressant medication(s) are eligible to participate.
* Inability to provide informed consent or complete any of the study tasks as determined by the principal investigator.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available to other researchers who contact the project Principal Investigator via email. Data will be available to such requests 1 year after the conclusion of recruitment.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year after the conclusion of recruitment
Access Criteria: Researchers should contact the project Principal Investigator via email.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 adult daily cigarette users completed a single laboratory session. We recruited non-treatment-seeking adults who use cigarettes daily to complete a single session utilizing a randomized, parallel design. We recruited individuals from the greater Philadelphia area using print and digital media advertisements.
Period: Overall Study
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Customized [Count of Participants; unit: Participants]
  ≥21 and ≤ 65 | 35 | 35 | 70
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at birth: Male | 22 | 22 | 44
  Sex at birth: Female | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 22 | 19 | 41
  Race: White or Caucasian | 11 | 15 | 26
  Race: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Smoking History Information_Past 7-day cigarettes per day [Mean (Standard Deviation); unit: Cigarettes] — During the study session, participants were asked to report on the number of cigarettes smoked in the past 7 days.
  Cigarettes | 13.6 (6.6) | 15.1 (7.6) | 14.4 (7.1)
Smoking History Information_Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: units on a scale] — At their study session, participants were asked to complete the Fagerstrom Test for Nicotine Dependence (FTND) measure, which assesses a Baseline level of Nicotine Dependence for cigarette smokers. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 4.6 (1.9) | 5.3 (2.2) | 4.9 (2.1)
Smoking History Information_Years Smoked [Mean (Standard Deviation); unit: Years] — During the study session, participants were asked to report on the total number of years they have smoked cigarettes.
  Years | 33.5 (11.5) | 32.1 (10.8) | 32.8 (11.1)
Smoking History_Type of Cigarette [Number; unit: Participants] — During the study session participants were asked to report the type of cigarette they smoked, menthol versus non-menthol.
  Participants
    Menthol | 24 | 25 | 49
    Non-Menthol | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Attention: Latency (Time Until First Fixation) for Image
Description: We defined areas of interest (AOIs) encompassing the image and text portions of each PWL. For each AOI, we examined attention measures of latency (time until the first fixation in the AOI; i.e., how quickly attention is drawn to the AOI), latency duration (length of the first fixation; i.e., how long the AOI is initially viewed), and total fixation time (sum of all fixations in the AOI; i.e., overall viewing allocation, accounting for viewing the same AOI multiple times). Analyses examined the mean of each outcome across the four PWLs within each condition.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 2612 (308) | 978 (313)

2. Primary Outcome: Attention: Latency (Time Until First Fixation) for Text
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 1001 (214) | 798 (218)

3. Primary Outcome: Attention: Latency Duration (Time of Fixation) for Image
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 160 (11) | 183 (13)

4. Primary Outcome: Attention: Latency Duration (Time of Fixation) for Text
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 150 (9) | 165 (9)

5. Primary Outcome: Attention: Total Fixation Time for Image
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 3532 (524) | 7887 (532)

6. Primary Outcome: Attention: Total Fixation Time for Text
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
ms | 4889 (436) | 3643 (443)

7. Primary Outcome: Recall: Participants Ability to Recall Condition Image
Description: Participants will view 11 warning label images and would be required to identify the warning label images they saw during their eye tracking portion of the session. This outcome measure (Recall -Image) was assessed in a percentage unit of measure. The percentages are not whole numbers for these items because it's the mean % correct for the condition, or the average percent correct across the four images for the group. The results in the Outcome Measure Data table demonstrate the percentage of participants who correctly identified the images from their condition (4 of the 11 images presented to participants were from their randomized condition; A or B).
Time Frame: Day 1
Measure: Mean (Standard Error); unit: percentage of correct images
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
percentage of correct images | 98.6 (1.0) | 95.7 (1.6)

8. Primary Outcome: Recall: Participants Ability to Recall Condition Text
Description: Participants will view 11 warning label text statements and would be required to identify the warning label text statements they saw during their eye tracking portion of the session. This outcome measure (Recall -Text) was assessed in a percentage unit of measure. The percentages are not whole numbers for these items because it's the mean % correct for the condition, or the average percent correct across the four images for the group. The results in the Outcome Measure Data table demonstrate the percentage of participants who correctly identified the text statements from their condition (4 of the 11 images presented to participants were from their randomized condition; A or B).
Time Frame: Day 1
Measure: Mean (Standard Error); unit: percentage of correct text
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
percentage of correct text | 82.9 (3.9) | 86.5 (3.1)

9. Primary Outcome: Knowledge of Smoking Harms
Description: All participants will select harms caused by tobacco from a list of health issues and diseases, before as well as after viewing the warning labels on the screen. Pre and post warning label exposure knowledge of smoking harms were assessed by using an exploratory scale that asked participants if cigarette smoking caused a list of 18 health conditions with a 5-point response scale, (1=definitely yes 2= probably yes, 3 = might or might not, 4 = probably not, 5 = definitely not).
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
Number analyzed (Participants) | 35 | 35
units on a scale
  Head and Neck Cancer | 1.4 (0.2) | 3.0 (0.2)
  Hearing Loss | 3.3 (0.2) | 3.9 (0.2)
  Lung Disease | 1.3 (0.1) | 1.3 (0.1)
  Vertigo | 3.0 (0.2) | 3.3 (0.2)
  Cataracts | 1.8 (0.2) | 3.4 (0.2)
  Depression | 2.7 (0.2) | 3.1 (0.2)
  Erectile Dysfunction | 3.2 (0.2) | 3.3 (0.2)
  Bladder Cancer | 1.9 (0.2) | 2.8 (0.2)
  Bloody Urine | 1.8 (0.2) | 3.5 (0.2)
  Harm to Children | 1.4 (0.1) | 1.5 (0.1)
  Blindness | 2.0 (0.2) | 3.5 (0.2)
  COPD (Chronic Obstructive Pulmonary Disease) | 1.6 (0.1) | 1.3 (0.1)
  Type II Diabetes | 2.0 (0.2) | 3.6 (0.2)
  Stunted Fetal Growth | 1.6 (0.1) | 1.5 (0.1)
  Heart Disease | 1.4 (0.1) | 1.5 (0.1)
  Stroke | 1.7 (0.1) | 1.9 (0.1)
  Macular Degeneration | 2.8 (0.2) | 3.0 (0.2)
  COVID-19 | 4.0 (0.2) | 4.1 (0.2)

ADVERSE EVENTS:
Time Frame: This is a single session study where adverse event data was not collected.
Arm/Group | Condition A (Lesser-known Harms) | Condition B (Well-known Harms)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Our small sample size and lack of variability in recall and post-exposure knowledge outcomes prevented exploring causal associations between these measures and attention outcomes. We operationalized "understanding" of harms as an increase in knowledge and used aided recall measures, which may have higher endorsement rates compared to unaided recall. other approaches to assessing these outcomes may yield different results and require further investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT04936724/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04936724/ICF_002.pdf